CLINICAL TRIAL: NCT02066844
Title: Phase II Study of Navigator vs Standard Needle Injection for Hip
Brief Title: Navigator vs Standard Needle Injection for Hip
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cartiva, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTC-0369
Record Dates: First submitted 2014-02-17; First posted 2014-02-20 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Hip Pain Etiology Unknown
Keywords: Hip Pain; Hip Injection; Hip Fracture; Hip Bursitis; Hip Arthritis; Hip Sciatica
MeSH Terms: conditions — Hip Fractures | interventions — Betamethasone; betamethasone sodium phosphate; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Manual Needle Injection (Active Comparator): 2cc of Celestone and 5cc of Lidocaine will be administered by the nurse or surgeon
  Interventions: Drug: Celestone; Drug: Lidocaine
- Navigator Injection (Experimental): 2cc of Celestone and 5cc of Lidocaine will be administered using the Navigator by the nurse or surgeon
  Interventions: Drug: Celestone; Drug: Lidocaine

INTERVENTIONS:
Drug: Celestone — 2cc
  Other Names: Betamethasone Sodium Phosphate
Drug: Lidocaine — 5cc

SUMMARY:
The purpose of this randomized, parallel-group, single-blinded, single center, Phase II study is to collect data to compare the comfort and patient satisfaction of a hip injection delivered via the Navigator compared to a standard needle injection. In addition, delivery preparation will be compared between a Navigator injection and a standard hip injection. The data collected from this pilot study will serve as the basis to design a larger multi-center study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ≥18 years of age, of any race or ethnicity;
* Capable of completing self-administered questionnaires;
* Patients with suspected intra-articular hip pain who have failed conservative care (conservative care defined as a standard regimen of home or outpatient physical therapy, activity modification, trial of at least one NSAID) for at least 3 months;
* Candidate for a hip injection;
* Have been informed of the nature of the study, agreeing to its requirements, and have signed the informed consent approved by the Institutional Review Board/Ethics Committee.
* Subjects are able to understand and speak English

Exclusion Criteria:

* History of intra-articular injection within the last 3 months prior to the injection procedure;
* Complex regional pain syndrome;
* History of prior hip surgery;
* History of substance abuse;
* Known history of hypersensitivity to local anesthetics of the amide type;
* Contraindicated for Celestone (betamethasone sodium phosphate);
* Contraindicated for Lidocaine Hydrochloride;
* Is a prisoner or ward of the state;
* Are unable to meet the treatment and follow up protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Injection Pain as measured by VAS for both treatment groups | From 1 week to 12 weeks post-injection

SECONDARY OUTCOMES:
Global Patient Satisfaction | From 1 week to 12 weeks post-injection
Drug Preparation Time | From 1 week to 12 weeks post-injection
Hip Pain and Function | From 1 week to 12 weeks post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Brian Giordano, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No